CLINICAL TRIAL: NCT06055101
Title: Intrathecal Bupivacaine-Dexmedetomidine Compared to Intrathecal Bupivacaine-Neostigmine in Elective Caesarean Sections, Randomized Clinical Trial
Brief Title: Regional Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reham Ali Abdelhaleem Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Reham Ali Abdelhaleem Abdelrahman, Anesthesia lecturer M.D., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AA-2023
Record Dates: First submitted 2023-08-30; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia, Obstetric
MeSH Terms: interventions — Dexmedetomidine; Neostigmine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DEXMEDETOMIDINE (Other): Group 1 ( 18 patients ) were received 10 mg (2ml) hyperbaric bupivacaine and 0.1 ml (10 μg) DXM and 0.1 ml normal saline.
  Interventions: Drug: DEXMEDETOMIDINE
- Neostigmine (Other): Group 2( 18 patients ) were received 10 mg (2ml) hyperbaric bupivacaine and 0.1 ml (50 μg) neostigmine and 0.1 ml normal saline.
  Interventions: Drug: Neostigmine
- Bupivacaine (Other): Group 3 ( 18 patients ) were received 10 mg (2ml) hyperbaric bupivacaine and 0.2 ml normal saline as control.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: DEXMEDETOMIDINE — DXM is a nonselective α2 agonist. Alpha2 adrenoreceptors, the overall response to α2 adrenoreceptors agonists is related to the stimulation of α2 adrenoreceptors located in the CNS and spinal cord. These receptors are involved in the sympatholysis, sedation, and antinociception effects of α2 adrenoreceptors.
  DEXMEDETOMIDINE (DXM) DXM shows a high ratio of specificity for the α2 receptor (α2/α11600: 1) compared with clonidine (α2/α1 200: 1), making it a complete α2 agonist. (76) DXM belongs to the imidazole subclass of α2 receptor agonists, similar to clonidine. It is freely soluble in water.
  Arms: DEXMEDETOMIDINE
Drug: Neostigmine — Neostigmine is an indirect cholinomimetic agent. It produces its primary effects by inhibiting the action of AChe, which hydrolyzes acetylcholine (ACh) to choline and acetic acid. By inhibiting AChe, the indirect-acting drug increases the concentration of spinal endogenous ACh. This drug is, in effect, amplifiers of endogenous ACh and act primarily where ACh is physiologically release. It combines reversibly with AChe by the formation of an ester linkage, which lasts about 30 minutes. The pharmacokinetic of neostigmine administered by bolus injection is linear with respect to bolus injection.
  Arms: Neostigmine
Drug: Bupivacaine — The onset of sensory blockade following spinal block with bupivacaine is very rapid (within one minute); maximum motor blockade and maximum dermatome level are achieved within 15 minutes in most cases.
  The conduction of nerve impulses along nerve fibers is related to changes in the electrical gradient across the nerve membrane and movement of predominantly sodium ions (but also potassium ions) from intracellular to extracellular fluid and vice versa. Bupivacaine work by reversibly blocking specific areas of the nerve cell membrane, known as sodium channels. It contains a mixture of ionized and un-ionized particles which, when injected into body tissues, make more un-ionized particles available, which are lipid soluble and able to penetrate the nerve cell membrane.
  Arms: Bupivacaine

SUMMARY:
Spinal anesthesia is an established technique used in obstetric surgeries, It provides adequate analgesia both intra and post-operative and also avoids complications associated with general anesthesia for mother and fetus. The quality of spinal anesthesia has been reported to be improved by using additives Dexmedetomidine is a highly selective α2-adrenoreceptor agonist that has been introduced to anesthesia. It produces dose-dependent sedation, anxiolysis, and analgesia without respiratory depression. Neostigmine is an anticholinesterase agent, which inhibits the hydrolysis of acetylcholine by competing with acetylcholine for attachment to acetyl cholinesterase; administration of Neostigmine through intrathecal route apparently activates the descending pain inhibitory system that relies on spinal cholinergic interneuron. Study conducted to evaluate whether neostigmine given by intrathecal route with 0.5% hyperbaric bupivacaine for spinal anesthesia can provide prolongation of sensory blockade duration as effective as dexmedetomidine given by the same route and in compination with same drug with lower cost, more stable hemodynamics and comparable side effects. After obtaining Institutional Ethics Committee approval and written informed consent,54 patients American Society of Anesthesiologist (ASA) physical status I and II were enrolled into the study and were randomlyassigned into 3 groups. Group 1were received 10 mg (2ml) hyperbaric bupivacaine and 0.1 ml (10 μg) DXM and 0.1 ml normal saline, Group 2 were received 10 mg (2ml) hyperbaric bupivacaine and 0.1 ml (50 μg) neostigmine and 0.1 ml normal saline and Group 3were received 10 mg (2ml) hyperbaric bupivacaine and 0.2 ml normal saline as control.

The investigators measured the time to reach T4 dermatome sensory block, peak sensory level, Time to reach Bromage 3 motor block, the regression time for sensory and motor block, also the investigators measured hemodynamic, sedation score, visual analogue score, any complications occurred and Apgar score for fetus during blockade and the investigators assessed the duration of pain relief .

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I and II patients
2. Age: 18 - 40 years
3. Height 150 - 170 cm
4. Weight 70 - 110 kg.

Exclusion Criteria:

1. Patient refusal
2. Cardiac diseases as ( ischemic heart disease, severe valvular stenosis, pulmonary hypertension, uncontrolled arrhythmias )
3. Severe labile hypertension BP more than 160 / 100 )
4. Raised intracranial pressure or pre-existing neurological disorders, such as multiple sclerosis.
5. Patients with coagulopathy: platelets < 100,000 INR ≥ 1.3 or therapeutic use of anti-coagulants.
6. Inability to communicate and understand the aim of the project.
7. Patients with history of allergic reaction to LA, DXM or Neostigmine.
8. Skin infection at injection site or systemic bacteremia.
9. Failure of the block and need for general anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Time started from the end of intrathecal injection till achievement of a bilateral sensory block at T10 | 90 seconds
  assessed by a pin prick needle from caudal to cephalic direction

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Ali Abdelrahman, Cairo, Egypt